CLINICAL TRIAL: NCT01134276
Title: Prospective Study on the Comparison Between the Clinicopathological Outcomes According to the Methods of Preoperative Biliary Drainage in Periampullary Cancers Causing Obstructive Jaundice
Brief Title: Comparison Between Internal and External Preoperative Biliary Drainage in Periampullary Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Whe Kim, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1001-047-307
Record Dates: First submitted 2010-05-04; First posted 2010-05-31 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Periampullary Cancers With Obstructive Jaundice; Pancreas Head Cancer; Bile Duct Cancer; Ampulla of Vater Cancer
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTBD (Active Comparator): biliary drainage : PTBD procedure for obstructive jaundice in patients with periampullary cancer
  Interventions: Procedure: biliary drainage
- ERBD (Active Comparator): biliary drainage : ERBD/ENBD procedure for obstructive jaundice in patients with periampullary cancer
  Interventions: Procedure: biliary drainage

INTERVENTIONS:
Procedure: biliary drainage — biliary drainage via PTBD or ERBD/ENBD

SUMMARY:
Preoperative biliary drainage methods include percutaneous transhepatic biliary drainage (PTBD), endoscopic nasobiliary drainage (ENBD), and endoscopic retrograde biliary drainage (ERBD). Endoscopic biliary drainages often induce peritumoral inflammation and it increase difficulties in determining a proper resection margin. The purpose of this study is to compare the clinicopathological outcomes according to the methods of preoperative biliary drainage in periampullary cancers causing obstructive jaundice, and to find out a proper biliary drainage method.

ELIGIBILITY:
Inclusion Criteria:

* patient who have periampullary tumors causing obstructive jaundice
* patient age: ≥20 and ≤85
* resectable state of disease
* no history of previous chemotherapy or radiotherapy
* patients without uncontrollable severe cardiovascular, respiratory disease
* Karnofsky performance scale ≥70
* informed consent

Exclusion Criteria:

* patients with distant metastasis or locally advanced disease with major vascular invasion
* duodenal cancer
* biliary drainage before randomization
* previous chemotherapy or radiotherapy
* uncontrollable active infection except cholangitis
* severe comorbid disease (cardiac, pulmonary, cerebrovascular)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] van der Gaag NA, de Castro SM, Rauws EA, Bruno MJ, van Eijck CH, Kuipers EJ, Gerritsen JJ, Rutten JP, Greve JW, Hesselink EJ, Klinkenbijl JH, Rinkes IH, Boerma D, Bonsing BA, van Laarhoven CJ, Kubben FJ, van der Harst E, Sosef MN, Bosscha K, de Hingh IH, Th de Wit L, van Delden OM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for periampullary tumors causing obstructive jaundice; DRainage vs. (direct) OPeration (DROP-trial). BMC Surg. 2007 Mar 12;7:3. doi: 10.1186/1471-2482-7-3. PMID 17352805
- [Background] Speer AG, Cotton PB, Russell RC, Mason RR, Hatfield AR, Leung JW, MacRae KD, Houghton J, Lennon CA. Randomised trial of endoscopic versus percutaneous stent insertion in malignant obstructive jaundice. Lancet. 1987 Jul 11;2(8550):57-62. doi: 10.1016/s0140-6736(87)92733-4. PMID 2439854
- [Background] Sewnath ME, Karsten TM, Prins MH, Rauws EJ, Obertop H, Gouma DJ. A meta-analysis on the efficacy of preoperative biliary drainage for tumors causing obstructive jaundice. Ann Surg. 2002 Jul;236(1):17-27. doi: 10.1097/00000658-200207000-00005. PMID 12131081
- [Background] Saiki S, Chijiiwa K, Komura M, Yamaguchi K, Kuroki S, Tanaka M. Preoperative internal biliary drainage is superior to external biliary drainage in liver regeneration and function after hepatectomy in obstructive jaundiced rats. Ann Surg. 1999 Nov;230(5):655-62. doi: 10.1097/00000658-199911000-00007. PMID 10561089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 211 patients underwent pancreatoduodenectomy after preoperative biliary drainage at Seoul National University Hospital.
Pre-assignment Details: 144 patients and 68 patients were intended to be treated with ERBD/ENBD and PTBD, respectively. Among 144 patients, 39 patients were switched to PTBD due to a procedure failure. Finally, 104 and 107 patients were treated with ERBD/ENBD and PTBD, respectively. Clinical outcomes were compared on the basis on the final drainage method
Groups:
- ERBD: biliary drainage : biliary drainage via ERBD/ENBD
- PTBD: biliary drainage : biliary drainage via PTBD
Period: Overall Study
Arm/Group | ERBD | PTBD
Started | 104 | 107
Completed | 104 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ERBD: final biliary drainage procedure: biliary drainage via ERBD/ENBD
- PTBD: final biliary drainage procedure : biliary drainage via PTBD
- Total: Total of all reporting groups
Arm/Group | ERBD | PTBD | Total
Number analyzed (Participants) | 104 | 107 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.6) | 63.5 (9.0) | 64.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 75
  Male | 71 | 65 | 136
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 104 | 107 | 211

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infectious Complications After Biliary Drainage
Description: at least 90 days after operation change in serum bilirubin cholangitis blood test (complete blood cell count, liver function test, CRP)
Time Frame: within 120 days after drainage
Measure: Number; unit: participants
Groups:
- PTBD: finial biliary drainage procedure: biliary drainage via PTBD
- ERBD: finial biliary drainage procedure: biliary drainage via ERBD or ENBD
Arm/Group | PTBD | ERBD
Number analyzed (Participants) | 107 | 104
participants | 11 | 5

2. Secondary Outcome: Change in Total Serum Bilirubin After Drainage
Description: Effect of reducing serum total bilirubin after drainage in terms of Daily diminution of bilirubin(mg/dL/day)
Time Frame: within 14 days after drainage
Measure: Mean (Standard Deviation); unit: mg/dL/day
Groups:
- PTBD: Final biliary drainage procedure: biliary drainage via PTBD
- ENBD/ERBD: Final biliary drainage procedure: biliary drainage via ENBD/ERBD
Arm/Group | PTBD | ENBD/ERBD
Number analyzed (Participants) | 107 | 104
mg/dL/day | 0.7 (0.5) | 0.6 (0.4)

3. Secondary Outcome: Total Hospital Cost During Admission After Biliary Drainage
Description: Total hospital cost during admission after Biliary Drainage in US dollars
Time Frame: during hospital stay for biliary drainage procedure
Measure: Mean (Standard Deviation); unit: thousands in US dollars
Arm/Group | PTBD | ERBD
Number analyzed (Participants) | 107 | 104
thousands in US dollars | 16.0 (5.9) | 17.0 (7.5)

ADVERSE EVENTS:
Time Frame: 7 days after procedure such as PTBD and ENBD/ERBD per Intervention
Groups:
- PTBD: final biliary drainage procedure: biliary drainage via PTBD
  Adverse event will be monitored by examination of clinic doctor in both in-patient and out-patient setting
- ERBD: final biliary drainage procedure: biliary drainage via ERBD/ENBD
  Adverse event will be monitored by examination of clinic doctor in both in-patient and out-patient setting
Arm/Group | PTBD | ERBD
Serious Adverse Events (participants affected / at risk) | 29/107 | 23/104
Other Adverse Events (participants affected / at risk) | 0/107 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTBD (N=107) | ERBD (N=104)
Bleeding (Blood and lymphatic system disorders) | 6 (6) | 3 (3) — procedure associated bleeding event after PTBD or ENBD/ERBD
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 17 (17) — Procedure associated pancreatitis after PTBD and ENBD/ERBD
Cholangitis (Gastrointestinal disorders) | 9 (9) | 5 (5) — Procedure associated cholangitis after PTBD and ENBD/ERBD
tube malfunction (Surgical and medical procedures) | 9 (9) | 7 (7) — tube malfunction which should be managed with additional procedure after PTBD and ENBD/ERBD
Bile peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0) — Procedure associated peritonitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No